CLINICAL TRIAL: NCT00519519
Title: Intravenous Infusion of High Dose Omeprazole Versus Regular Dose Omeprazole on Recurrent Bleeding After Endoscopic Treatment of Bleeding Peptic Ulcers
Brief Title: Optimal Dose of Omeprazole After Endoscopic Treatment of Bleeding Peptic Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 78:10/03-098
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Bleeding Peptic Ulcers Disease
Keywords: Rebleeding after endoscopic therapy
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Active Comparator): regular dose versus high dose
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — intravenous 80mg bolus followed by 8mg / hr for 3 days
  Other Names: intravenous 40 mg om for 3 days

SUMMARY:
Bleeding peptic ulcers are one of the major causes of morbidity and mortality for hospital emergency admissions.The initial treatment is endoscopic therapy followed by intravenous omeprazole. However the optimal dosage of omeprazole is not known. We conducted this study to find out the optimal dosage in such clinical scenario.

DETAILED DESCRIPTION:
Introduction

Peptic ulcer bleeding (PUB) is a common and life threatening condition. Intravenous infusion of high dose omeprazole (80mg as bolus followed by 8 mg/hr for 72 hours ie 652 mg/72 hrs) after endoscopic therapy resulted in greater reductions of re-bleeding than did placebo. Thus the above regime became our departmental protocol. However, there is some evidence that both high dose and a regular dose of omeprazole (40mg once a day followed by a saline infusion ie 120mg/72 hrs) would be equally effective. We calculated that high dose regimen is about S$ 500 more expensive. The aim of our study is to determine the equivalence of both regimes in preventing re-bleeding rate (primary end-point), surgery and mortality in PUB patients.

Study design This is a single institution prospective randomized double-blind study. All patient with PUB (Forrest classification I, IIa and IIb: spurting or oozing bleeding, visible vessels and clot) had endoscopic treatments (adrenaline injection and/or heater probe). After successful endoscopic hemostasis, patients are randomized to receive a high or regular dose of omeprazole infusion. After 72 hours, both groups of patients are given oral omeprazole 40mg daily for 4 weeks. All patients are evaluated at the clinic at the end of 4 weeks. The primary end-point is rebleeding. Other secondary endpoints measured are surgery, duration of hospital stay and death.

ELIGIBILITY:
Inclusion Criteria:

1. Above 21 year old
2. OGD done within 48 hrs of admission
3. No recent upper GIT surgery past one month
4. Forrest Type I, IIa & IIb ulcer (Type Ia: Spurting, Ib:Oozing, IIa: Visible vessel, IIb: Clot)
5. Non-malignant ulcer
6. Informed consent taken

Exclusion Criteria:

1. Impaired hepatic function
2. Pregnancy
3. Lactation
4. Concomitant medication (warfarin, diazepam, phenytoin, chlarithromycin, cimetidine and digoxin)
5. Underlying malignancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-07; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Re-bleeding rate after endoscopic treatment of bleeding peptic ulcers | 30 days after endoscopic therapy

SECONDARY OUTCOMES:
Surgery, Death and Length of hospital stay | 30 days after endoscopic thearpy

CONTACTS AND LOCATIONS:
Overall Officials: Weng Hoong Chan, MBBS, FRCS, Principal Investigator — Singapore General Hospital; Weng Hoong Chan, MBBS, FRCS, Principal Investigator — Department of Surgery, Singapore General Hospital
Locations (4):
- Singapore (4):
  - Department of Surgery, Singapore General Hospital, Outram Road, Singapore, Outram Road
  - Singapore General Hospital, Outram Road, Singapore, Outram Road
  - Department of Surgery, Singapore General Hospital, Singapore, Outram Road
  - Singapore General Hospital, Singapore, Outram Road

REFERENCES:
- [Derived] Chan WH, Khin LW, Chung YF, Goh YC, Ong HS, Wong WK. Randomized controlled trial of standard versus high-dose intravenous omeprazole after endoscopic therapy in high-risk patients with acute peptic ulcer bleeding. Br J Surg. 2011 May;98(5):640-4. doi: 10.1002/bjs.7420. Epub 2011 Feb 8. PMID 21305536